CLINICAL TRIAL: NCT05615025
Title: Influence of Sevoflurane and Propofol on Maximum Muscular Strength, Speed of Contraction and Relaxation, in Humans: A Pilot Study
Brief Title: Influence of Sevoflurane and Propofol on Maximum Muscular Strength, Speed of Contraction and Relaxation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Denis SCHMARTZ, Anesthesiologists, Université Libre de Bruxelles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CHUB-ITF sevo-propofol
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Anesthesia, General; Neuromuscular Transmission Disorders
MeSH Terms: conditions — Neuromuscular Junction Diseases | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sevoflurane arm (Experimental): In this arm, anesthesia will be maintained by sevoflurane.
  Interventions: Drug: Sevoflurane
- Propofol arm (Experimental): In this arm, anesthesia will be maintained by propofol.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane — Anesthesia will be maintained by sevoflurane.
  Arms: Sevoflurane arm
Drug: Propofol — Anesthesia will be maintained by propofol.
  Arms: Propofol arm

SUMMARY:
Many drugs have an influence on neuromuscular transmission. In clinical practice, neuromuscular blocking agents are commonly used, but even in the absence of neuromuscular blocking agents, anesthetic drugs can influence neuromuscular transmission. Especially volatile anesthetic agents have a clinical impact on neuromuscular transmission, they have been shown to prolong and deepen the effect of neuromuscular blocking agents. But even in the absence of neuromuscular blocking agents, volatile anesthetics can impair neuromuscular transmission. One mechanism of action is the desensitization of the acetylcholine receptors by shifting them from a normal to a desensitized state. This effect can weaken neuromuscular transmission by reducing the margin of safety that normally exists at the neuromuscular junction, or can cause an apparent increase in the capacity of neuromuscular blocking agents to block transmission.

In this study, the influence of sevoflurane and propofol on the maximum force, maximum speed of contraction and relaxation will be measured at the adductor pollicis in patients having general anesthesia without the use of neuromuscular blocking agents. Maximum force and speed of contraction and relaxation will be measured before and after anesthesia by either sevoflurane or propofol. Primary outcome is the influence of either anesthetic agent on maximum muscular force and speed of contraction - relaxation, and if this influence is greater for volatile anesthetic agents than for intravenous anesthetic agents.

ELIGIBILITY:
Inclusion criteria

* Patients (male or female) from 18 - 80 years
* Scheduled for surgery without the use of neuromuscular blocking agents
* Health care insurance in Belgium
* Written informed consent

Exclusion Criteria:

* Any pathology involving neuromuscular transmission
* Confirmed neuropathy of any origin
* Expected anesthesia duration < 30 min
* Renal insufficiency defined as a glomerular filtration rate < 40 mL/min/m2
* Hepatic insufficiency defined as an increase > 1.5 * normal value of hepatic enzymes
* Confirmed or suspected pregnancy
* Language barrier
* Any patient which will receive unplanned neuromuscular blocking agents during surgery
* Any history of personal or familial suspected malignant hyperthermia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Maximum force at the adductor pollicis | 3 hours
  Maximum force developed by a voluntary contraction of the adductor pollicis will be measured during isometric contraction. Maximum force developped before and after anesthesia will be compared. The difference in force (Newton) will be measured.
Maximum speed of contraction at the adductor pollicis | 3 hours
  Maximum speed of contraction developed by a voluntary contraction of the adductor pollicis will be measured during isometric contraction. Maximum speed of contraction developped before and after anesthesia will be compared. The difference in force (Newton/seconds) will be measured.
Maximum speed of relaxation at the adductor pollicis | 3 hours
  Maximum speed of relaxation developed by a voluntary contraction of the adductor pollicis will be measured during isometric contraction. Maximum speed of relaxation developped before and after anesthesia will be compared. The difference in force (Newton/seconds) will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baurain MJ, Hoton F, D'Hollander AA, Cantraine FR. Is recovery of neuromuscular transmission complete after the use of neostigmine to antagonize block produced by rocuronium, vecuronium, atracurium and pancuronium? Br J Anaesth. 1996 Oct;77(4):496-9. doi: 10.1093/bja/77.4.496. PMID 8942335
- [Background] Chung F, Chan VW, Ong D. A post-anesthetic discharge scoring system for home readiness after ambulatory surgery. J Clin Anesth. 1995 Sep;7(6):500-6. doi: 10.1016/0952-8180(95)00130-a. PMID 8534468
- [Background] Debaene B, Frasca D, Moreillon F, D'Hollander AA. 100 Hz-5 s tetanic stimulation to illustrate the presence of "residual paralysis" co-existing with accelerometric 0.90 train-of-four ratio-A proof-of-concept study. Anaesth Crit Care Pain Med. 2021 Aug;40(4):100903. doi: 10.1016/j.accpm.2021.100903. Epub 2021 Jun 17. PMID 34147687
- [Background] Dubois PE, Mitchell J, Regnier M, Passeraub PA, Moreillon F, d'Hollander AA. The interest of 100 versus 200 Hz tetanic stimulations to quantify low levels of residual neuromuscular blockade with mechanomyography: a pilot study. J Clin Monit Comput. 2022 Aug;36(4):1131-1137. doi: 10.1007/s10877-021-00745-6. Epub 2021 Jul 24. PMID 34302578
- [Background] Feldman S, Karalliedde L. Drug interactions with neuromuscular blockers. Drug Saf. 1996 Oct;15(4):261-73. doi: 10.2165/00002018-199615040-00004. PMID 8905251
- [Background] Gage PW. Ion channels and postsynaptic potentials. Biophys Chem. 1988 Feb;29(1-2):95-101. doi: 10.1016/0301-4622(88)87028-5. PMID 2451942
- [Background] Karis JH, Gissen AJ, Nastuk WL. The effect of volatile anesthetic agents on neuromuscular transmission. Anesthesiology. 1967 Jan-Feb;28(1):128-34. doi: 10.1097/00000542-196701000-00014. No abstract available. PMID 6017421
- [Background] Ochiai R, Guthrie RD, Motoyama EK. Effects of varying concentrations of halothane on the activity of the genioglossus, intercostals, and diaphragm in cats: an electromyographic study. Anesthesiology. 1989 May;70(5):812-6. doi: 10.1097/00000542-198905000-00018. PMID 2719316
- [Background] Ochiai R, Guthrie RD, Motoyama EK. Differential sensitivity to halothane anesthesia of the genioglossus, intercostals, and diaphragm in kittens. Anesth Analg. 1992 Mar;74(3):338-44. doi: 10.1213/00000539-199203000-00004. PMID 1539811
- [Background] Pereda AE, Faber DS. Activity-dependent short-term enhancement of intercellular coupling. J Neurosci. 1996 Feb 1;16(3):983-92. doi: 10.1523/JNEUROSCI.16-03-00983.1996. PMID 8558267
- [Background] Raines DE. Anesthetic and nonanesthetic halogenated volatile compounds have dissimilar activities on nicotinic acetylcholine receptor desensitization kinetics. Anesthesiology. 1996 Mar;84(3):663-71. doi: 10.1097/00000542-199603000-00022. PMID 8659795
- [Background] Silverman DG, Brull SJ. The effect of a tetanic stimulus on the response to subsequent tetanic stimulation. Anesth Analg. 1993 Jun;76(6):1284-7. doi: 10.1213/00000539-199376060-00017. PMID 8098919
- [Background] Simons JC, Pierce E, Diaz-Gil D, Malviya SA, Meyer MJ, Timm FP, Stokholm JB, Rosow CE, Kacmarek RM, Eikermann M. Effects of Depth of Propofol and Sevoflurane Anesthesia on Upper Airway Collapsibility, Respiratory Genioglossus Activation, and Breathing in Healthy Volunteers. Anesthesiology. 2016 Sep;125(3):525-34. doi: 10.1097/ALN.0000000000001225. PMID 27404221
- [Background] Stauble CG, Stauble RB, Schaller SJ, Unterbuchner C, Fink H, Blobner M. Effects of single-shot and steady-state propofol anaesthesia on rocuronium dose-response relationship: a randomised trial. Acta Anaesthesiol Scand. 2015 Aug;59(7):902-11. doi: 10.1111/aas.12523. Epub 2015 May 12. PMID 25962311
- [Background] Tassonyi E, Charpantier E, Muller D, Dumont L, Bertrand D. The role of nicotinic acetylcholine receptors in the mechanisms of anesthesia. Brain Res Bull. 2002 Jan 15;57(2):133-50. doi: 10.1016/s0361-9230(01)00740-7. PMID 11849819
- [Background] Yamaoka K, Vogel SM, Seyama I. Na+ channel pharmacology and molecular mechanisms of gating. Curr Pharm Des. 2006;12(4):429-42. doi: 10.2174/138161206775474468. PMID 16472137